CLINICAL TRIAL: NCT01315886
Title: Conversion From Fast Acting Oral Opioids to Abstral® (SL Fentanyl) in Opioid Tolerant Cancer Patients With Breakthrough Pain
Brief Title: Conversion From Fast Acting Oral Opioids to Abstral®
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Orexo AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX20-005; 2010-020239-38 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Pain
Keywords: sublingual; fentanyl; titration; conversion; breakthrough cancer pain; pain intensity difference; PID; Edmonton Symptom Assessment System; ESAS
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SL Fentanyl conversion (Experimental): * Baseline period: 7-15 episodes of breakthrough cancer pain treated with prior IR opioid medication
  * Treatment period: Conversion to SL Fentanyl at a Fentanyl:Prior opioid conversion factor of 1:50 (using the estimated Morphine Sulphate Equivalent dose for the prior opioid). SL Fentanyl use was followed for 8-15 episodes of breakthrough cancer pain. SL Fentanyl dose could be titrated between episodes.
  Interventions: Drug: SL fentanyl

INTERVENTIONS:
Drug: SL fentanyl — SL fentanyl will be administered during 7- 15 BTcP episodes during a maximum period of 21 days, following a baseline period with standard BTcP treatment. The start dose of SL fentanyl is selected individually according to a standardized conversion ratio. The maximum start dose is limited to 400 μg. For a single BTcP episode no more than two (2) tablets or a maximum dose of 800 μg should be given.
  Other Names: Abstral

SUMMARY:
The purpose of this study is to evaluate safety and efficacy when using a novel dose conversion strategy to switch from immediate release oral opioids to sublingual (SL) fentanyl (Abstral) for treatment of breakthrough cancer pain (BTcP).

DETAILED DESCRIPTION:
The study aims to show that in the advanced stage of cancer the individual patient already on high doses of BTcP medication will benefit from starting treatment on a higher first dose of SL fentanyl thus reducing the number of dosing steps with insufficient pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained.
* 18 years or older, of both genders.
* Opioid tolerant patients
* Estimated frequency of BTcP 0.5-4 times a day.

Exclusion Criteria:

* Treatment with SL fentanyl within two weeks prior to screening.
* Recent or planned therapy that would alter pain or responses to analgesics.
* Treatment with monoamine oxidase inhibitor < 14 days before or concurrent with SL fentanyl treatment.
* Significantly reduced liver and/or kidney function.
* Significant prior history of substance abuse.
* Pregnancy, breast feeding or woman of childbearing potential not using adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-02-21 (Actual); Primary Completion 2011-12-07 (Actual); Study Completion 2011-12-07 (Actual)

PRIMARY OUTCOMES:
Response rate in patients converted to SL fentanyl. | 30 minutes post dose
  A subject is defined as responder if the change of Pain Intensity (PI) on the Numerical Rating Scale (NRS) rated from 0 to 10, at 30 minutes (PID30) is similar or higher after the conversion to SL fentanyl compared to baseline PID30 as assessed by standard care rescue treatment of BTcP episodes.

SECONDARY OUTCOMES:
Responder rate in patients converted to SL fentanyl as assessed by the PID15. | 15 minutes post dose
Edmonton Symptom Assessment System (ESAS) Symptom Distress Score (SDS) | 24 hour assessment on days with pain episodes
Patient's global assessment of treatment (patient satisfaction). | 2 occasions
Patients preference of treatment (baseline treatment/SL fentanyl). | end of study
Occurrence of AEs, withdrawals | during a maximum treatment period of 21 days.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Pettersson, MD, PhD, Study Chair — Orexo AB
Locations (1):
- Smärtavdelning B42, Anestesikliniken Karolinska University Hospital, Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No